CLINICAL TRIAL: NCT06339164
Title: Breech Delivery Skills. Formal Lecture vs Digital Learning in Resident Learning Program.
Brief Title: Breech Delivery Skills. Resident Learning Program
Acronym: Breech
Status: Not yet recruiting | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Claudio Celentano, MD, G. d'Annunzio University
Other Study IDs: ObGynEASC006
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Breech Presentation; Before Labor
Keywords: breech, learning, mannequin
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Formal lecture: residents undergoing frontal lecture one month before the scenario
  Interventions: Other: skills and learning quality in breech delivery
- Digital learning: residents learning digitally the topic for at least one month before the scenario
  Interventions: Other: skills and learning quality in breech delivery

INTERVENTIONS:
Other: skills and learning quality in breech delivery — evaluation of different skill retention and learning quality after different learning methods

SUMMARY:
Breech delivery is one of the mail topic in emergency obstetrics for Italian Board of Obstetrics and Gynecology. Formal frontal lecture and digital learning represent nowadays the two typical learning methods. A bedside evaluation it's not feasible due to rarity of such emergency, due to the common senior physicians involvement when it occurs, and due to medico-legal risks. Mannequin scenario represents the best way of skill evaluation

DETAILED DESCRIPTION:
Residents will be recruited for "breech delivery" in two different ways. One group (20) will attend a formal frontal lecture on breech delivery of at least one hour. A second group matched for sex distribution, age, residency year (20) will receive a digital lecture. After one month the two groups will test their abilities on a low fidelity mannequin. The simulation session will be recorded and evaluated by 5 specialists in a blind way. During the simulation the main topics of breech extraction are recorded. All residents will receive a questionnaire identifying the subject, previous experience bedside or in a course, and the agreement for video recording and data analysis. After the simulation test they will receive a second questionnaire indicating improvement levels (using a Kirkpatrick model and a 5-point Likert scale).

ELIGIBILITY:
Inclusion Criteria: residents in University of Chieti Medical school -

Exclusion Criteria: none

-

Ages: 24 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all residents undergoing lecture for obstetric emergencies
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Skills capacities | 1 months
  Skills at the scenario (maneuvers). Deriving form charts recorded during the scenario and time enalpsed
Skills capacities | 1 month
  Skills at the scenario evaluated for 5 supervisors

SECONDARY OUTCOMES:
learning qualities | 1 month
  from questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Celentano, Pescara, PE, Italy

IPD SHARING:
Plan to Share IPD: No
questionnaire on Goggle forms